CLINICAL TRIAL: NCT03965559
Title: The Efficacy of Plasmapheresis and Double Filtration Plasmapheresis (DFPP) in Kidney Transplant Patients With Suspected Rejection: A Retrospective Study
Brief Title: The Efficacy of Plasmapheresis and Double Filtration Plasmapheresis (DFPP) in Kidney Transplant
Status: Completed | Type: Observational
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kajohnsak Noppakun, Assistant Professor, Chiang Mai University
Other Study IDs: MED-2558-03579
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Kidney Transplant Rejection; Plasmapheresis; Kidney Replacement
MeSH Terms: interventions — Plasmapheresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- plasmapheresis group: Kidney transplant patients who had been diagnosed or suspected of graft rejection and underwent the plasmapheresis during January 2006 to October 2015
  Interventions: Procedure: plasmapheresis
- double filtration plasmapheresis (DFPP) group: Kidney transplant patients who had been diagnosed or suspected of graft rejection and underwent the double filtration plasmapheresis (DFPP) during January 2006 to October 2015
  Interventions: Procedure: plasmapheresis

INTERVENTIONS:
Procedure: plasmapheresis — Plasmapheresis is the removal, treatment, and return or exchange of blood plasma or components thereof from and to the blood circulation. It is thus an extracorporeal therapy (a medical procedure performed outside the body).[Wikipedia]
  DFPP is a selectively removal of the immunoglobulin fraction from the serum and, as a result, to minimize the volume of substitution fluid required. [Tanabe K. Double-filtration plasmapheresis. Transplantation. 2007 Dec 27;84(12 Suppl):S30-2.]
  Other Names: double filtration plasmapheresis (DFPP)

SUMMARY:
At present, the number of end-stage kidney disease patients is increasing. Kidney transplant surgery is one of the treatments that give patients a better survival rate than hemodialysis or abdominal dialysis. In Thailand, there were 5,729 kidney transplant patients or 88.9 cases per million population in 2012. Among this number, 465 were new surgical patients or 7.2 cases per million population.

From the year 2007-2012, the survival rate of the kidney donor from living donor kidney transplant (LDKT) was 98.5 percent and 93.3 percent at 1 and 5 years, respectively.

The most common cause of graft loss was chronic rejection by 33% of all graft loss. However, 16.1 percent were unknown reasons for graft loss.

The research question is "In patients with kidney transplantation who suspected graft rejection" Is it true that doing plasmapheresis or DFPP is no different.

The researcher therefore conducted a comparative study. Is plasmapheresis or DFPP effective or different side effects?

DETAILED DESCRIPTION:
Rejection condition can be divided into 2 groups, namely cellular rejection and antibody-mediated rejection (AbMR) by acute AbMR treatment according to the guidelines for care for kidney transplant patients in Thailand, 2014. The introduction of a single filter plasma (plasmapheresis) or 2 filters (DFPP) in combination with IVIG (intravenous immunoglobulin), which may or may not be given methylprednisolone. If the patients did not response to the treatment, Rituximab or Bortezomib was considered.

Only one previous study showed that among 29 graft rejected patients treated with plasmapheresis, 37.9% had subsequently graft loss and the rest of them had significantly decreasing creatinine level at 1 month follow-up. Another group of 10 graft rejected patients treated with DFPP, 40% had subsequently graft loss. Six patients had decreasing creatinine level at 1 month follow-up.

Both groups do not have complications or side effects from plasmapheresis or DFPP.

The researcher therefore conducted a comparative study.

Is plasmapheresis or DFPP effective or different side effects in treating post-kidney transplant patients who suspected of graft rejection?

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 15 years
* Kidney transplant patients who have been diagnosed or suspected of having graft rejection from antibodies

Exclusion Criteria:

* Incomplete data

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The research team will search for medical records, outpatients and / or inpatients of the index cases of kidney transplant patients who had been diagnosed or suspected of graft rejection and was treated with either plasmapheresis or DFPP during January 2006 to October 2015
  To record the following details
  * Demographic data of patients (Demographic Data)
  * Clinical clinical presentation
  * Existing diseases and medications
  * Kidney transplantation information Landscape used Levels of autoimmune conditions during the 6 months before renal salivation
  * Preliminary laboratory results Including sugar levels Blood fat level Before treatment and after treatment at 1 week, 1 month and 3 months
  * Renal biopsy results before and after treatment (if any)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Treatment response | 1 week
  Compare treatment response rates after complete treatment with plasmapheresis and DFPP
Treatment response | 1 month
  Compare treatment response rates after complete treatment with plasmapheresis and DFPP
Treatment response | 3 month
  Compare treatment response rates after complete treatment with plasmapheresis and DFPP

SECONDARY OUTCOMES:
Kidney loss | 1 week, 1 month, and 3 month
  Comparison of kidney loss rate at 1 week, 1 month and 3 months after complete treatment during plasmapheresis with DFPP
Complications | 1 week, 1 month, and 3 month
  Compare the rate of occurrence, side effects and complications during treatment plasmapheresis and DFPP

CONTACTS AND LOCATIONS:
Overall Officials: Kajohnsak Noppakun, MD, Principal Investigator — Chiang Mai University

IPD SHARING:
Plan to Share IPD: No
If it is asked for or requested for

REFERENCES:
- [Background] Noppakun K, Ingsathit A, Pongskul C, Premasthian N, Avihingsanon Y, Lumpaopong A, Vareesangthip K, Sumethkul V; Subcommittee for Kidney Transplant Registry; Thai Transplantation Society. A 25-year experience of kidney transplantation in Thailand: report from the Thai Transplant Registry. Nephrology (Carlton). 2015 Mar;20(3):177-83. doi: 10.1111/nep.12378. PMID 25492162
- [Background] Westall GP, Paraskeva MA, Snell GI. Antibody-mediated rejection. Curr Opin Organ Transplant. 2015 Oct;20(5):492-7. doi: 10.1097/MOT.0000000000000235. PMID 26262460
- [Background] Kirubakaran MG, Disney AP, Norman J, Pugsley DJ, Mathew TH. A controlled trial of plasmapheresis in the treatment of renal allograft rejection. Transplantation. 1981 Aug;32(2):164-5. doi: 10.1097/00007890-198108000-00019. No abstract available. PMID 7027553
- [Background] Allen NH, Dyer P, Geoghegan T, Harris K, Lee HA, Slapak M. Plasma exchange in acute renal allograft rejection. A controlled trial. Transplantation. 1983 May;35(5):425-8. doi: 10.1097/00007890-198305000-00006. PMID 6342220
- [Background] Bonomini V, Vangelista A, Frasca GM, Di Felice A, Liviano D'Arcangelo G. Effects of plasmapheresis in renal transplant rejection. A controlled study. Trans Am Soc Artif Intern Organs. 1985;31:698-703. No abstract available. PMID 3915622
- [Background] Brown CM, Abraham KA, O'Kelly P, Conlon PJ, Walshe JJ. Long-term experience of plasmapheresis in antibody-mediated rejection in renal transplantation. Transplant Proc. 2009 Nov;41(9):3690-2. doi: 10.1016/j.transproceed.2009.06.197. PMID 19917368
- [Background] Larpparisuth N, Vongwiwatana A, Vareesangthip K, Cheunsuchon B, Parichatikanon P, Premasathian N. Clinicopathologic features and treatment response of early acute antibody-mediated rejection in Thai kidney transplant recipients: a single-center experience. Transplant Proc. 2014;46(2):474-6. doi: 10.1016/j.transproceed.2013.12.022. PMID 24655992
- [Background] Larpparisuth N, Premasathian N, Vareesangthip K, Cheunsuchon B, Parichatikanon P, Vongwiwatana A. Clinicopathologic characteristics and outcomes of late acute antibody-mediated rejection in Thai kidney transplant recipients: a single-center experience. Transplant Proc. 2014;46(2):477-80. doi: 10.1016/j.transproceed.2014.01.003. PMID 24655993
- [Background] Gungor O, Sen S, Kircelli F, Yilmaz M, Sarsik B, Ozkahya M, Hoscoskun C, Ok E, Toz H. Plasmapheresis therapy in renal transplant patients: five-year experience. Transplant Proc. 2011 Apr;43(3):853-7. doi: 10.1016/j.transproceed.2011.03.025. PMID 21486614
- [Background] Haas M, Sis B, Racusen LC, Solez K, Glotz D, Colvin RB, Castro MC, David DS, David-Neto E, Bagnasco SM, Cendales LC, Cornell LD, Demetris AJ, Drachenberg CB, Farver CF, Farris AB 3rd, Gibson IW, Kraus E, Liapis H, Loupy A, Nickeleit V, Randhawa P, Rodriguez ER, Rush D, Smith RN, Tan CD, Wallace WD, Mengel M; Banff meeting report writing committee. Banff 2013 meeting report: inclusion of c4d-negative antibody-mediated rejection and antibody-associated arterial lesions. Am J Transplant. 2014 Feb;14(2):272-83. doi: 10.1111/ajt.12590. PMID 24472190